CLINICAL TRIAL: NCT04840862
Title: Impact of Rifabutin on the Pharmacokinetics of Elexacaftor/Tezacaftor/Ivacaftor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Paul Beringer, Professor of Clinical Pharmacy, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-21-00315
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — elexacaftor, ivacaftor, tezacaftor drug combination; Rifabutin

STUDY DESIGN:
Intervention Model Description: A single group of subjects will receive a single dose of trikafta (orange tablet) in period 1. After washout period greater or equal to 2 days, subjects will receive 300 mg/d of rifabutin on day 1 through 17 and a single dose of trikafta (orange tablet) on day 15 in period 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- rifabutin (Experimental): Rifabutin PO [two 150mg capsules] ; Trikafta PO [one orange tablet containing ELX 100mg, TEZ 50mg, and IVA 75mg]
  Interventions: Drug: Trikafta [orange tablet containing ELX 100mg, TEZ 50mg, and IVA 75mg]; Drug: Rifabutin 300mg

INTERVENTIONS:
Drug: Trikafta [orange tablet containing ELX 100mg, TEZ 50mg, and IVA 75mg] — Subjects will receive a single dose of trikafta (orange tablet) on day 1 of period 1 and on day 15 of period 2.
Drug: Rifabutin 300mg — After washout period greater or equal to 2 days, subjects will receive 300 mg/d of rifabutin on days 1 through 17 of period 2.

SUMMARY:
This is a prospective, single-center, fixed-sequence, nonrandomized, open-label study in healthy adults to investigate the impact of rifabutin on the pharmacokinetics of trikafta.

DETAILED DESCRIPTION:
Trikafta (Elexacaftor [ELX], Tezacaftor [TEZ], Ivacaftor[IVA]) is contraindicated with concomitant use of strong inducers as co-administration of rifampin decreased the area-under-the concentration time curve (AUC) of IVA by 89%, creating a therapeutic challenge to the treatment of non-tuberculosis mycobacteria (NTM) infection in people with cystic fibrosis (CF). While rifabutin also induces CYP3A4 activity, its effects appear to be more moderate when compared with rifampin. Therefore, we hypothesize that rifabutin can be co-administered with an adjusted dose of ELX/TEZ/IVA in patients being treated for NTM pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign informed consent prior to any study-related activities.
* Male or female participants between 18 and 65 years of age inclusive.
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination findings, and clinical laboratory test results
* Body mass index (BMI) of 17.5 to 30.5 kg/m2, inclusive; and a total body weight >50kg (110 lbs).
* Willing to stop using any herbal or natural health products for 2 weeks prior to and during the study including: Grapefruit, grapefruit juice, St. John's Wort.
* Participant must use a reliable method of birth control while they are participating in the study; for instance an intrauterine device (IUD), condom with spermicidal gel or foam, diaphragm with spermicidal gel or foam, vasectomy, tubal ligation, hysterectomy or abstinence or female must be post-menopausal for at least one year.

Exclusion Criteria:

* Female subjects of childbearing potential with positive urine pregnancy test at screening.
* Female subjects who are breastfeeding.
* Use of CYP3A modulators (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin, azole drugs, telithromycin, clarithromycin, erythromycin)
* Any significant acute or chronic medical illness that might confound the results of the study or pose an additional risk in administrating study drugs to the subject, as determined by the investigator.
* Any condition that could affect drug absorption (eg, gastrectomy, pancreatitis).
* Any major surgery within 4 weeks of study drug administration.
* Blood donation of approximately 1 pint (500 mL) within 56 days before study drug administration.
* Known hypersensitivity to rifamycins
* Patients with hepatic impairment (Child-Pugh Class B or C) and/or with history of hepatobiliary disease or liver function test elevations.
* Renal insufficiency (eGFR < 60 mL/min)
* History of uveitis and/or current eye or vision problems with the exception of corrective lenses.
* Contact lens use during study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
24h area-under the plasma concentration time curve (AUC) of ELX/TEZ/IVA in the absence and the presence of concomitant rifabutin | 22 days
  To assess the impact of rifabutin on the AUC of ELX/TEZ/IVA

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ELX/TEZ/IVA in the absence and the presence of concomitant rifabutin | 22 days
  To assess the impact of rifabutin on the Cmax of ELX/TEZ/IVA

CONTACTS AND LOCATIONS:
Overall Officials: Adupa P Rao, M.D., Study Director — Keck Medicine of USC
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Sanders M, Hong E, Chung PS, Rao AP, Cohn W, Beringer P. Evaluation of the drug interaction between rifabutin and elexacaftor/tezacaftor/ivacaftor (ETI). J Cyst Fibros. 2026 Jan;25(1):151-157. doi: 10.1016/j.jcf.2025.09.002. Epub 2025 Sep 16. PMID 40957819